CLINICAL TRIAL: NCT04177316
Title: Differential Hypermethylation Status of the VTRNA2-1 Promoter in Hepatocellular Carcinoma as an Independent Factor After Partial Hepatectomy
Brief Title: Hypermethylation of VTRNA2-1 Promoter in HCC Outcome
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201801969B0
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Hepatocellular Carcinoma Resectable
Keywords: VTRNA2-1 promoter; recurrence; methylation
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — frozen specimen of tumor and normal parts at Central Biobank of Chang Gung Memorial Hospital
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypermethylation: The hypermethylation group was defined as differential methylation status of tumor- normal ≥ 5%.
- hypomethylation/no change: The hypomethylation were defined as differential methylation status of tumor- normal <5%

SUMMARY:
The clinic-pathological data were retrieved from the cancer registry database from the Cancer Center of Chang Gung Memorial Hospital, Linkou branch. Of the 92 HCC patients with partial hepatectomies enrolled. The biological specimen was studied with approval.

DETAILED DESCRIPTION:
This study was approved by the Institute Review Board (IRB) of Chang Gung Memorial Hospital, Linkou Branch (IRB 201801969B0). The clinic-pathological data were retrieved from the cancer registry database from the Cancer Center of Chang Gung Memorial Hospital, Linkou branch. Of the 92 HCC patients with partial hepatectomies enrolled, all patients had curative hepatectomy and those with different cancers were excluded. HCC tumor tissue and normal tissue, 3 cm from the tumor margin, were stored immediately in a -80 degree freezer at the Central Biobank of Chang Gung Memorial Hospital. The personal information was protected with decoding and registered with number.

ELIGIBILITY:
Inclusion Criteria:

subjects with pathologic diagnosis of hepatocellular carcinoma curative partial hepatectomies

Exclusion Criteria:

history of different malignant disease. subjects cannot be treated with curative surgery.

Ages: 20 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: HCC patients with curative partial hepatectomies and the pathology reports proved.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
disease free survival (DFS) | a month
  The length of time from curative hepatectomies treatment and recurrence or mortality

SECONDARY OUTCOMES:
Overall survival | a month
  The length of time from hepatectomies treatment for HCC and still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chin Yu, MD, PhD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Ming-Chin Yu, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No